CLINICAL TRIAL: NCT06026735
Title: Comprehensive Profiling of Promising Biomarkers in Exosomes From Non-small Cell Lung Cancer With Central Nervous System Metastasis
Brief Title: Non-small Cell Lung Cancer With Central Nervous System Metastasis
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202209032RINB
Record Dates: First submitted 2022-10-25; First posted 2023-09-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-08

CONDITIONS: Lung Cancer With Central Nervous System Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- lung cancer with brain metastasis
  Interventions: Other: lung cancer with brain /leptomeningeal metastasis
- lung cancer with leptomeningeal metastasis
  Interventions: Other: lung cancer with brain /leptomeningeal metastasis

INTERVENTIONS:
Other: lung cancer with brain /leptomeningeal metastasis — Cerebrospinal fluid was obtained from the cerebrospinal cavity of non-small cell lung cancer patients with central nervous system metastasis, blood was obtained from veins, and metastatic lung cancer tumor tissue was obtained from surgically resected brain tumors or meningeal tumors. Then comprehensively analyze the exosomes contained in the aforementioned samples, and compare and analyze the clinical data of the patients, so as to explore whether the cancer cell-related substances contained in the cerebrospinal fluid, blood and tumor tissue can be used to predict lung cancer metastasis and Bioindicators of treatment effect.

SUMMARY:
Cerebrospinal fluid was obtained from the cerebrospinal cavity of non-small cell lung cancer patients with central nervous system metastasis, blood was obtained from veins, and metastatic lung cancer tumor tissue was obtained from surgically resected brain tumors or meningeal tumors. Then comprehensively analyze the exosomes contained in the aforementioned samples, and compare and analyze the clinical data of the patients, so as to explore whether the cancer cell-related substances contained in the cerebrospinal fluid, blood and tumor tissue can be used to predict lung cancer metastasis and Bioindicators of treatment effect.

ELIGIBILITY:
Inclusion Criteria:

- A. Non-small cell lung cancer patients diagnosed with brain metastases or meningeal metastases on brain computed tomography (CT) or magnetic resonance (MRI) images.

B. Patients with non-small cell lung cancer who are about to undergo surgical brain surgery, such as brain tumor resection, lumbar abdominal drainage, Euclidean storage, or ventriculoperitoneal drainage.

Exclusion Criteria:

- A. Non-small cell lung cancer patients without brain metastases or meningeal metastases.

B. Physical condition does not allow surgical removal of the tumor.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-small cell lung cancer patients with brain metastases or meningeal metastases.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-01-13 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
predict lung cancer metastasis and Bioindicators of treatment effect | follow 3 years
  Cerebrospinal fluid was obtained from the cerebrospinal cavity of non-small cell lung cancer patients with central nervous system metastasis, blood was obtained from veins, and metastatic lung cancer tumor tissue was obtained from surgically resected brain tumors or meningeal tumors. Then comprehensively analyze the exosomes contained in the aforementioned samples, and compare and analyze the clinical data of the patients, so as to explore whether the cancer cell-related substances contained in the cerebrospinal fluid, blood and tumor tissue can be used to predict lung cancer metastasis and Bioindicators of treatment effect.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan